CLINICAL TRIAL: NCT00539448
Title: Phase IV, Open Label, Non-comparative, Multi-center, Study of the Effects of Both Insulin Glargine & Insulin Glulisine in Type I Diabetes Mellitus Patients.
Brief Title: Gulf, Lantus, Apidra Evaluation in Type 1 Diabetics Study
Acronym: GLANS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Medical Affairs Study Director, sanofi-aventis
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LANTU_L_01578
Record Dates: First submitted 2007-10-03; First posted 2007-10-04 (Estimated); Last update posted 2009-09-25 (Estimated); Status verified 2009-09

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin Glargine; insulin glulisine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): combination of insulin Glargine & insulin Glulisine as basal bolus regimen
  Interventions: Drug: insulin glargine; Drug: insulin glulisine

INTERVENTIONS:
Drug: insulin glargine — in combination with insulin Glulisine as bolus regimen
Drug: insulin glulisine — in combination with insulin Glargine as bolus regimen

SUMMARY:
Primary objective :

To evaluate the efficacy (in terms of change in HbA1c readings starting from baseline then after 13 weeks & at the end of the study which will be after 26 weeks) in subjects with type I diabetes mellitus.

Secondary objective :

* Recording the average daily dose of both insulin Glulisine & insulin Glargine in type I DM.
* Recording adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed type I diabetic patients
* Type I diabetes treated with basal-bolus regimen including 3 or more injections of Regular Human Insulin per day
* BMI, 26-40 kg/m2
* HbA1c, 7.5%-10%
* Median 2Hrs post -prandial more than or equal to 140 mg/dl (more than or equal to 7.8 mmol/L)
* FPG more than or equal to 120 mg/dl (more than or equal to 6.7 mmol/L)
* Willingness to accept, and ability to inject insulin Glargine therapy

Exclusion Criteria:

* Pregnancy : The use of LANTUS & APIDRA during pregnancy is not contraindicated. However, in the absence of supportive data, Sanofi- Aventis Pharmaceuticals cannot specifically recommend the use of Lantus in this patient population

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 98 (Actual)
Dates: Start 2007-04; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Evaluating the Glycemic control of the regimen : Change in A1C levels | from baseline to study end

SECONDARY OUTCOMES:
Average daily dose : - For both insulin Glulisine & insulin Glargine. - FBG and PPBG if possible ? | from baseline to study end

CONTACTS AND LOCATIONS:
Overall Officials: Hisham - MAHMOUD, MD, Study Director — Sanofi
Locations (4):
- Sanofi-aventis administrative office, Manama, Bahrain
- Sanofi-aventis administrative office, Kuwait City, Kuwait
- Sanofi-Aventis Administrative Office, Doha, Qatar
- Sanofi-aventis administrative office, Dubai, United Arab Emirates